CLINICAL TRIAL: NCT01861912
Title: Arsenic Trioxide TACE and Intravenous Administration Compared With Arsenic Trioxide TACE Alone in Unresectable Hepatocellular Carcinoma: a Randomized, Parallel, Controlled, Multi-center Clinical Study
Brief Title: Arsenic Trioxide TACE and Intravenous Administration in Unresectable Hepatocellular Carcinoma
Acronym: ACTION
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Ligong Lu, MD, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDREC2013109H(R1)
Record Dates: First submitted 2013-05-16; First posted 2013-05-24 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma, Hepatocellular; Arsenic trioxide
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Ethiodized Oil; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arsenic trioxide TACE (Active Comparator): Arsenic trioxide TACE: arsenic trioxide powder 20mg dissolved in lipiodol(the dosage of lipiodol is decided according to the volume of the target lesion)is used for transcatheter arterial chemoembolization(TACE). TACE will be repeated after 4~6 weeks if it is necessary according to the assessment from imaging modalities.
  Interventions: Device: Arsenic trioxide TACE; Drug: lipiodol
- Arsenic trioxide TACE+IV (Experimental): 1. Arsenic trioxide TACE: arsenic trioxide powder 20mg dissolved in lipiodol(the dosage of lipiodol is decided according to the volume of the target lesion)is used for transcatheter arterial chemoembolization(TACE). TACE will be repeated after 4~6 weeks if it is necessary according to the assessment from imaging modalities.
  2. Arsenic trioxide intravenous infusion: arsenic trioxide powder 0.15mg/Kg/d(maxim 10mg/d) dissolved in 250ml 0.9% sodium chloride solution is used for intravenous infusion.Every course will last for 3 weeks and the next course will be continued after 1 week suspension.Intravenous infusion will be suspended 3 days before and 7~14 days after TACE.
  Interventions: Device: Arsenic trioxide TACE; Drug: Arsenic trioxide intravenous infusion; Drug: lipiodol; Drug: NaCl solution

INTERVENTIONS:
Device: Arsenic trioxide TACE — Arsenic trioxide powder 20mg dissolved in lipiodol(the dosage of lipiodol is decided according to the volume of the target lesion)is used for transcatheter arterial chemoembolization(TACE). TACE will be repeated after 4~6 weeks if it is necessary according to the assessment from imaging modalities
Drug: Arsenic trioxide intravenous infusion — Arsenic trioxide intravenous infusion: arsenic trioxide powder 0.15mg/Kg/d(maxim 10mg/d) dissolved in 250ml 0.9%NaCl solution is used for intravenous infusion.Every course will last for 3 weeks and the next course will be continued after 1 week suspension.Intravenous infusion will be suspended 3 days before and 7~14 days after TACE.
  Arms: Arsenic trioxide TACE+IV
Drug: lipiodol — Lipiodol is used to dissolve arsenic trioxide for TACE,with the dosage decided according to the volume of the target lesion.
Drug: NaCl solution — 250ml NaCl solution is used to dissolve the arsenic trioxide for intravenous infusion.
  Arms: Arsenic trioxide TACE+IV

SUMMARY:
The purpose of this study is to determine whether compared with arsenic trioxide TACE alone, arsenic trioxide TACE and intravenous administration could further prolong the overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent;
* Histological or clinical diagnosis of hepatocellular carcinoma（HCC）;
* The target lesion should had at least one diameter line available for measurement, with the maximum diameter ≥5cm and ≤10cm；
* Barcelona Clinic Liver Cancer staging B or C;
* Child-Pugh liver function class: score≤7；
* Eastern Cooperative Oncology Group performance 0 or 1;
* At least 12 weeks life expectancy;
* Never received systemic treatment, such as oral molecularly targeted drugs and systemic chemotherapy;
* Be able to abide by the treatment and follow-up plan；
* Adequate results for laboratory tests, including:

  1. Neutrophil count≥1.5×109/L, platelet count≥60×109 /L; hemoglobin≥85g/L;
  2. Total bilirubin≤51.3 μmol/L, albumin≥28 g/L,and alanine aminotransferase and aspartate aminotransferase≤5 times the upper limit of the normal range;
  3. Amylase and lipase≤1.5 times the upper limit of the normal range
  4. Serum creatinine≤20 g/L
  5. Prothrombin time international normalized ratio ≤1.7; or prothrombin time≤4seconds above control;
  6. Left ventricular ejection fraction≥50% according to two-dimensional echocardiography;
* Contraception: during the trail and 12 weeks after the withdrawal, female of childbearing age (WOCBP), WOCBP whose male partners receive study drug or male must use appropriate contraceptive to avoid pregnancy;

Exclusion Criteria:

* Disease should be excluded:

  1. CT / MRI showed diffuse lesions;
  2. Extrahepatic metastasis (metastasis in lungs not included);
  3. Invasion in the main portal vein / vena cava or other major vascular;
  4. Previous shunt surgery;
  5. PreviousTACE or transarterial embolization for HCC, unless there is a untreated lesion;
  6. Hepatic encephalopathy in the past or present;
  7. Current ascites requiring treatment;
* Medical history and concomitant diseases:

  1. Previous or current cancer other than HCC, unless it is cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis and T1). Cancer having received curative treatment 5 years ago will not be excluded;
  2. Disease history in the cardiovascular system as the following:

  (a)Uncontrolled hypertension；(b)Congestive heart failure in New York Heart Association grade 3 or 4; (c)Active coronary artery disease within 12 months, unstable angina or newly diagnosed angina/myocardial infarction;(d)Arrhythmia requiring drugs other than β-blockers and digoxin;(e)Valvular heart disease ≥ CTCAE grade 2； c) Corrected QT interval (Fridericia)> 450 ms confirmed by 2 ECGs in a row d) Thrombotic or embolic events within 6 months, e) Gastrointestinal bleeding within 6 months; f) Unstable and / or active stomach ulcer within 6 months, unless gastroscopy showed it to be fully recovered; g) Variceal bleeding within 6 months; h) Unhealed wound or ulcer, fracture within 3 months; i) Major surgery, open biopsy, or severe trauma within 3 weeks; j) History of organ transplant or subjects in the transplant waiting list; k) Uncontrolled abnormal thyroid function; l) HIV infection; m) Active or untreated hepatitis B;
* laboratory tests unsuitable for the enrollment：

  1. Hyponatremia, serum sodium <130 mmol / L；
  2. Hypokalemia, serum potassium <3.5 mmol / L；
* Allergic reactions to arsenic trioxide and any other drugs used in this trail;
* Forbidden therapies and/or drugs:

  1. Condensation treatment (e.g., warfarin or heparin);
  2. Chronic antiplatelet therapy (Aspirin ≥ 300 mg / day; clopidogrel ≥ 75 mg / day);
  3. Radiotherapy within 4 weeks;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time to Progression | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  Time to progression in our study is defined as the time from a patient's enrollment to the time for disease progression (according to Recist1.1).

SECONDARY OUTCOMES:
Overall Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  Overall survival in our study is defined as the time from a patient's enrollment to the time for death.
Quality of Life | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  Quality of life is assessed according to the FACT-Hep questionnaire.
Safety | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  Safety of our treatment plan will be assessed according to the Common Terminology Criteria for Adverse Events（CTCAE） 3.0

OTHER OUTCOMES:
Extrahepatic Metastasis Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  Extrahepatic metastasis rate is defined as the proportion of the extrahepatic metastasis for patients who were absent of extrahepatic metastasis at enrollment.
Recurrence Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  Recurrence rate is defined as the proportion of the recurrence in the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ligong Lu, Doctor, Principal Investigator — Guangdong Provincial People's Hospital